CLINICAL TRIAL: NCT02045069
Title: A Phase II/III, Randomized, Placebo Controlled Trial of Efficacy and Safety of Ivermectin in Children and Adult Patients With Dengue Infection
Brief Title: Efficacy and Safety of Ivermectin Against Dengue Infection
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Collaborators: Ministry of Health, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESIDEN
Record Dates: First submitted 2014-01-13; First posted 2014-01-24 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 days Ivermectin (Experimental): Ivermectin 200 - 400 µg/kg once daily for 2 days
  Interventions: Drug: 2 days Ivermectin
- 3 days Ivermectin (Experimental): Ivermectin 200-400 µg/kg once daily for 3 days
  Interventions: Drug: 3 days Ivermectin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 2 days Ivermectin — 200-400 µg/kg once daily for 2 days and placebo once daily at D3
  Other Names: Mectizan; Ivomec; Stromectol
  Arms: 2 days Ivermectin
Drug: 3 days Ivermectin — 200 -400 µg/kg once daily for 3 days
  Arms: 3 days Ivermectin
Drug: Placebo — Placebo once daily for 3 days
  Arms: Placebo

SUMMARY:
This is a Phase II/III, Randomized, Double-Blind, Placebo-Controlled Study of Efficacy and Safety of Ivermectin in Children and Adult patients with Dengue Infection.

DETAILED DESCRIPTION:
Patients with confirmed dengue infection who meet all inclusion and exclusion criteria will be enrolled in the study and admitted in the hospital. Patients will be randomly assigned in a pre-specified ratio of 1:1:1 to one of the following study groups: ivermectin 200-400 µg/kg single daily dose for 2 days, ivermectin 200-400 µg/kg single daily dose for 3 days, or placebo. Tablets of ivermectin or placebo will be administered for 3 days. Clinical exam will be performed daily during hospitalization and blood samples will be collected for hematology, clinical chemistry, serology, viral load and quantitative nonstructural 1 (NS1) antigen. Safety assessment will be conducted during admission. Patients will be discharged one day after fever subsidence and will be asked to return 2 weeks after first dose of study medication for safety assessment and blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages of 15 or greater.
* History or presence of fever (temperature > 38°C) of ≤ 72 hr duration.
* Clinical suspicion of dengue infection such as high fever without an evidence or suspected focus of infection on clinical examination.
* Positive NS 1 strip assay

Exclusion Criteria:

* Clinically significant abnormal laboratory results which are deemed to be unassociated with dengue infection
* Clinical evidence or a history of significant respiratory, metabolic, renal, hepatic, hematologic or chronic diseases
* History of autoimmune, immune dysfunction disorder or taking warfarin
* Clinical suspicion of any bacterial infection
* Pregnancy and lactating women

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Time to resolution of viremia | Every 12 hr, from date of randomization until resolution of viremia or until fever subsides for 1 day, whichever came first.

SECONDARY OUTCOMES:
Time to clearance of NS1 antigen | Every 12 hr, from date of randomization until resolution of viremia or until fever subsides for 1 day, whichever came first.
Time of subsidence of fever | From date of randomization until fever subsides

CONTACTS AND LOCATIONS:
Overall Officials: Panisadee Avirutnan, MD, PhD., Principal Investigator — Division of Dengue Hemorrhagic Fever Research Department of Research and Development, Faculty of Medicine Siriraj Hospital Mahidol University, Bangkok 10700, THAILAND
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Ooi EE. Repurposing Ivermectin as an Anti-dengue Drug. Clin Infect Dis. 2021 May 18;72(10):e594-e595. doi: 10.1093/cid/ciaa1341. No abstract available. PMID 33124646